CLINICAL TRIAL: NCT06384508
Title: The Effectiveness of a Virtual Reality Intervention on Trauma-related Shame in Sexually Abused Adolescents: A Single-case Experimental Study
Brief Title: Decrease Trauma-related Shame With Virtual Reality: The Effectiveness of SHINE-VR
Acronym: SHINE-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Collaborators: University of Amsterdam (Other)
Responsible Party: Principal Investigator, Carlijn Bergwerff, Associate Professor, Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL83340.058.23
Record Dates: First submitted 2024-03-01; First posted 2024-04-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Shame
Keywords: shame; sexual abuse; virtual reality; self-compassion

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design (ABC) with two different baseline lengths
Who Masked: Participant
Masking Description: The participants are unaware of different baseline lengths
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHINE-VR Baseline 1 week (Active Comparator): Participants will receive SHINE-VR additionally to regular trauma treatment. The baseline phase starts after trauma processing, e.g. after module 6 of TF-CBT or processing of the traumatic event with EMDR.
  This group has a one week baseline, 3 weeks intervention, and 2 week follow-up phase.
  Interventions: Behavioral: SHINE-VR
- SHINE-VR Baseline 2 weeks (Active Comparator): Participants will receive SHINE-VR additionally to regular trauma treatment. The baseline phase starts after trauma processing, e.g. after module 6 of TF-CBT or processing of the traumatic event with EMDR.
  This group has a two week baseline, 3 weeks intervention, and a 1 week follow-up phase.
  Interventions: Behavioral: SHINE-VR

INTERVENTIONS:
Behavioral: SHINE-VR — The SHINE-VR takes place after trauma processing, e.g. after module 6 of TF-CBT or processing of the traumatic event with EMDR, and is followed by the rest of the regular treatment. SHINE-VR consists of the following 3 VR sessions à 45min:
  * Introduction: getting acquainted with VR, playing a VR game developed for the feasibility study (Krupljanin et al., in preparation), receiving psychoeducation about seeking help.
  * Shame: virtual group therapy setting, psychoeducation about shame, virtual peers sharing thoughts of shame and their learnings/positive affirmations.
  * Self-compassion: practicing self-compassion using an immersive perspective-changing task in VR.

SUMMARY:
Suffering from PTSD in childhood can have detrimental formative consequences. Researchers have been eager to develop effective interventions and to enhance treatment motivation since the introduction of the diagnosis of PTSD in the DSM. With evolving understanding of the disorder, its definition and criteria have changed over the course of time. The most recent change involves the addition of the criterium D of negative affects or emotions in relation to PTSD, the feeling of shame amongst others. Individuals experiencing interpersonal trauma, such as sexual abuse, are at high-risk developing trauma-related shame, which in turn can impact the course and effectiveness of PTSD treatment. Shame-inducing situations are typically being avoided, and the feelings are not disclosed to peers and other people. Hence, acknowledging and sharing feelings of shame as well as practicing self-compassion have been proposed to reduce the impact of that negative self-conscious emotion. These aspects get partially tackled in evidence-based trauma therapies, however, there appears to be a need for a more specific trauma-related shame intervention in addition to existing treatments. Recent research has focused on developing such interventions for adults and has reported positive effects.

To our knowledge, there is no intervention specifically tackling trauma-related shame in adolescents. Virtual Reality (VR) is a promising tool for such an intervention. Findings suggest that including VR in a treatment results in high treatment satisfaction and that it is highly motivating for its users, which is a crucial component for treatment success.

The goal of this study is to test the effectiveness of a short-term VR shame intervention (SHINE-VR) for adolescents suffering from PTSD after having experienced sexual abuse. The primary objectives of this study to assess the effect of SHINE-VR on trauma-related shame, self-compassion, and PTSD symptom reduction, to investigate whether treatment motivation, an increase in self-compassion, and a decrease in trauma-related shame are associated with PTSD symptom reduction.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 17 years old at inclusion
* Interpersonal trauma (sexual abuse); in case of multiple traumas the main trauma should be sexual abuse
* Indication for PTSD treatment
* Getting trauma treatment as usual
* Adequate command of the Dutch language

Exclusion Criteria:

* Known mental disability
* Epilepsy

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Trauma-related shame | Daily throughout the 6 weeks, resulting in 42 assessments
  Shame experienced in relation to sexual abuse will be measured with a self-developed questionnaire. The first 4 items are based on the Dutch translation of the Shame and Guilt After Trauma Scale. Each item is rated on a 5-point Likert scale. Higher scores mean worse outcome. 2 items are reversed. Higher scores mean worse outcome.
Self-compassion | Daily throughout the 6 weeks, resulting in 42 assessments
  Self-compassion will be measured with the Dutch translation of the Self-Compassion Scale-Youth version. Each of the 6 items is rated on a 1-5 Likert scale, 3 of them are reversed. The outcome measure is the sum score of all items divided by the number of items. Higher scores mean better outcome.

SECONDARY OUTCOMES:
PTSD symptoms | Daily on weekdays throughout the 6 weeks, resulting in 30 assessments
  PTSD symptoms will be measured with the Kind en Jeugd Traumascreener. Items 1-20 measuring the symptoms will be used, each item is rated on a 0-3 Likert scale. The outcome measure is the sum score of all items. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - GGZ Delfland, The Hague, Haaglanden
  - iMindU Practice for Child, Adolescent and Adult Psychiatry, Leiden, South Holland
  - LEVVEL, Amsterdam
  - Kenter Jeugdhulp, Haarlem
  - LUMC Curium, Oegstgeest

IPD SHARING:
Plan to Share IPD: Yes
Identifiable information of the participants will be encrypted for the further processing and analyzing of the corresponding data. Once the project is completed and the paper(s) has been published, the encryption key and the personal data will be deleted. Following paragraph from the template of the Institute of Education and Child Studies will be used:
  I consent to my and my child's participation in the study (Title Research) I also give permission to store and use the pseudonymised research data about me and my child that is collected in this research and to share it with other researchers if necessary.
Supporting Information: Study Protocol, SAP
Time Frame: We will store the data according to the University regulations on data management of projects assessed by the Medical Ethical committee, allowing the data to be FAIR for at least 15 years after publication.
Access Criteria: A CC-BY license will be used. Since sensitive data will be collected, it will only be shared with researchers upon request. Requests for information will be reviewed by the first and last author.
URL: https://dataverse.nl/

REFERENCES:
- [Result] Aakvaag HF, Thoresen S, Wentzel-Larsen T, Dyb G, Roysamb E, Olff M. Broken and guilty since it happened: A population study of trauma-related shame and guilt after violence and sexual abuse. J Affect Disord. 2016 Nov 1;204:16-23. doi: 10.1016/j.jad.2016.06.004. Epub 2016 Jun 11. PMID 27318595
- [Result] Neff KD, Bluth K, Toth-Kiraly I, Davidson O, Knox MC, Williamson Z, Costigan A. Development and Validation of the Self-Compassion Scale for Youth. J Pers Assess. 2021 Jan-Feb;103(1):92-105. doi: 10.1080/00223891.2020.1729774. Epub 2020 Mar 3. PMID 32125190
- [Result] Sachser C, Berliner L, Risch E, Rosner R, Birkeland MS, Eilers R, Hafstad GS, Pfeiffer E, Plener PL, Jensen TK. The child and Adolescent Trauma Screen 2 (CATS-2) - validation of an instrument to measure DSM-5 and ICD-11 PTSD and complex PTSD in children and adolescents. Eur J Psychotraumatol. 2022 Aug 1;13(2):2105580. doi: 10.1080/20008066.2022.2105580. eCollection 2022. PMID 35928521
- [Result] Drieschner KH, Boomsma A. Validation of the Treatment Motivation Scales for Forensic outpatient treatment (TMS-F). Assessment. 2008 Jun;15(2):242-55. doi: 10.1177/1073191107311651. Epub 2008 Feb 1. PMID 18245208